CLINICAL TRIAL: NCT06302231
Title: Effects of Time-restricted Eating Combined With Aerobic Exercise Training on Body Composition and Cardiometabolic Parameters in Women With Overweight and Obesity: a Randomized Clinical Trial
Brief Title: Effects of Time-restricted Eating and Aerobic Exercise Training in Women With Overweight and Obesity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Alvaro Reischak-Oliveira, Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16690919.5.0000.5347
Record Dates: First submitted 2024-02-19; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Time Restricted Eating; Obesity; Intermittent Fasting; Overweight and Obesity; Time Restricted Feeding
MeSH Terms: conditions — Intermittent Fasting; Obesity; Overweight | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Time-Restricted Eating and Aerobic Exercise Performed in Fasted State (Experimental): Participants will be prescribed a diet plan to promote weight loss, but no food will be provided to them.
  Diets will be formulated to contain 50% energy as carbohydrate, 20% as protein, and 30 % as fat.
  Participants will be instructed to divide their daily energy intake between three meals each day (lunch, afternoon snack, and dinner).
  Participants will be instructed to eat from 12.00 until 20.00 (8-hour window). Aerobic exercise sessions will be carried out during the morning shift with participants in a fasted state.
  Interventions: Behavioral: Dietary and Exercise Approaches
- Time-Restricted Eating and Aerobic Exercise Performed in Fed State (Active Comparator): Participants will be prescribed a diet plan to promote weight loss, but no food will be provided to them.
  Diets will be formulated to contain 50% energy as carbohydrate, 20% as protein, and 30 % as fat.
  Participants will be instructed to divide their daily energy intake between three meals each day (lunch, afternoon snack, and dinner).
  Participants will be instructed to eat from 12.00 until 20.00 (8-hour window). Aerobic exercise sessions will be carried out during the afternoon shift with participants in a fed state.
  Interventions: Behavioral: Dietary and Exercise Approaches
- Time-Restricted Eating (Other): Participants will be prescribed a diet plan to promote weight loss, but no food will be provided to them.
  Diets will be formulated to contain 50% energy as carbohydrate, 20% as protein, and 30 % as fat.
  Participants will be instructed to divide their daily energy intake between three meals each day (lunch, afternoon snack, and dinner).
  Participants will be instructed to eat from 12.00 until 20.00 (8-hour window). Participants in this arm will not perform aerobic exercise training.
  Interventions: Behavioral: Dietary Approach

INTERVENTIONS:
Behavioral: Dietary and Exercise Approaches — Intermittent fasting plus energy restriction combined with aerobic exercise performed in a fasted state.
  Arms: Time-Restricted Eating and Aerobic Exercise Performed in Fasted State
Behavioral: Dietary and Exercise Approaches — Intermittent fasting plus energy restriction combined with aerobic exercise performed in a fed state.
  Arms: Time-Restricted Eating and Aerobic Exercise Performed in Fed State
Behavioral: Dietary Approach — Intermittent fasting plus energy restriction without aerobic exercise training.
  Arms: Time-Restricted Eating

SUMMARY:
Time-restricted eating (TRE) is a dietary approach that aims to increase fasting time and decrease the eating window. Promising TRE effects on weight loss and improvements in some cardiometabolic risk factors have been reported in studies in animals and humans. However, the impacts of TRE combined with aerobic exercise training in individuals with overweight and obesity have been insufficiently investigated.

Additionally, aerobic training performed in a fasted state appears to promote physiological adaptations that may improve the metabolic health in individuals with overweight and obesity.

The present study investigates the effects of 8 weeks of TRE associated with aerobic training in a fasted state versus a fed state on body composition and cardiometabolic parameters in women with overweight and grade 1 obesity.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Body mass index (BMI) between 25 and 34.9 kg/m²;
* Age between 20 and 40 years;
* Not engaged in any structured exercise program;
* Weight stable for ~3 months before the beginning of the study;
* Able to give written informed consent.

Exclusion Criteria:

* Current smoker;
* Habitual drinkers (>1 serving/day) of alcoholic beverages;
* Cardiometabolic diseases (dyslipidemia, diabetes, hypertension, etc);
* Current treatment with medication or supplements which significantly affect the main studied variables;
* Bariatric surgery;
* Night-shift workers;
* Strict vegetarian/vegan;
* Pregnancy, planned pregnancy (within the study period), lactating;
* Postmenopausal women;
* Self-reported menstrual cycle irregularities;
* Habitual fasting window >16 hours;
* Concomitant participation in other studies.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity (indices) | Change from baseline. Measured at baseline and after 8 weeks.
  Including but not limited to the Sensitivity Matsuda index

SECONDARY OUTCOMES:
Insulin resistance (indices) | Change from baseline. Measured at baseline and after 8 weeks.
  Including but not limited to Homeostatic Model Assessment for Insulin Resistance (HOMA-IR).
Fasting insulin levels (µIU/mL) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by enzyme-Linked Immunosorbent Assay
Fasting glucose levels (mg/dL) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by colorimetric method
Glucose tolerance | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by oral glucose tolerance test (2-h OGTT)
Fasting lipid profile levels | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by colorimetric method
β cell function (indices) | Change from baseline. Measured at baseline and after 8 weeks.
  Including but not limited to HOMA-β
Fat Mass (kg) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by Dual-energy X-ray Absorptiometry under fasting condition.
Fat Percentage (%) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by Dual-energy X-ray Absorptiometry under fasting condition.
Fat Free Mass (kg) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by Dual-energy X-ray Absorptiometry under fasting condition.
Body Weight (kg) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by Dual-energy X-ray Absorptiometry under fasting condition.
Body Weight (kg) | Change from baseline. Measured at baseline and after 4, and 8 weeks.
  Measured on a digital scale.
Bone Mineral Content (kg) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by Dual-energy X-ray Absorptiometry under fasting condition.
Body Mass Index (kg/m^2) | Change from baseline. Measured at baseline and after 8 weeks.
  Calculated from weight in kilograms divided by height in meters squared.
Fasting ketones (β-hydroxybutyrate) levels (mmol/L) | Change from baseline. Measured at baseline and after 8 weeks.
Resting metabolic rate (Kcal/day) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by indirect calorimetry under resting and fasting conditions.
Substrate Oxidation (respiratory exchange ratio) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by indirect calorimetry under resting and fasting conditions.
Absolute Peak oxygen consumption | Change from baseline. Measured at baseline and after 4, and 8 weeks.
  Measured by an open-circuit spirometry system. Absolute value expressed in litres of oxygen per minute (L/min).
Relative Peak oxygen consumption | Change from baseline. Measured at baseline and after 4, and 8 weeks.
  Measured by an open-circuit spirometry system. Relative to body weight and expressed in milliliters of oxygen per minute (mL/kg/min).
Fasting Leptin Levels | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by enzyme-Linked Immunosorbent Assay
Fasting Adiponectin Levels | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by enzyme-Linked Immunosorbent Assay
Inflammatory Markers Levels | Change from baseline. Measured at baseline and after 8 weeks.
  Including but not limited to TNF-α (tumor necrosis factor-alpha) and IL-10 (Interleukin-10); Measured by enzyme-Linked Immunosorbent Assay
LDL-cholesterol levels | Change from baseline. Measured at baseline and after 8 weeks.
  Measured using the Friedewald equation.
Non-HDL-cholesterol levels | Change from baseline. Measured at baseline and after 8 weeks.
  Calculated as total cholesterol minus HDL-cholesterol.